CLINICAL TRIAL: NCT01865591
Title: A Clinical Trial for the Assessment of Safety and Efficacy of the UltraSOUND Mediated InTerVentional Treatment of Resistant Hypertension
Brief Title: Feasibility Study of Renal Denervation for the Treatment of Resistant Hypertension
Acronym: SoundITV
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sound Interventions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SITV-CL-0001
Record Dates: First submitted 2013-05-23; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension; uncontrolled hypertension; resistant hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal denervation (Experimental): Subjects are treated with unfocussed ultrasound-based renal denervation and are maintained on baseline anti-hypertensive medications.
  Interventions: Device: Ultrasound-based Renal Denervation

INTERVENTIONS:
Device: Ultrasound-based Renal Denervation
  Other Names: Sound TX System

SUMMARY:
The aim of this study is to assess the potential therapeutic benefit of catheter-based renal sympathetic denervation using therapeutic unfocussed ultrasound in a single-arm feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled hypertension (defined as SBP ≥ 140 mmHg during 24Hr Ambulatory BP monitoring)
* Current treatment with ≥ 3 anti-hypertensive drugs (including at least one diuretic)
* Renal artery diameter ≥5mm by digital angiography
* Accessibility of renal vasculature

Exclusion Criteria:

* Estimated GFR < 45
* Type 1 Diabetes
* Known renovascular abnormalities (eg, renal artery stenosis, previous renal artery stenting or angioplasty)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | 30 days
  All cause death, renal artery occlusion, renal artery stenosis, renal infarction and/or renal failure

SECONDARY OUTCOMES:
Change from baseline in office blood pressure measurement | 30 days, 3 months, 6 months, 9 months, 12 months
Change from baseline in ambulatory 24-hour blood pressure measurement | 6 months, 12 months
Change from baseline in renal artery dimensions | 30 days
  Change in renal artery dimensions as measured by renal angiography, CT, or MRI
Change from baseline in creatinine | 6 months
Adverse events and device complications | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia